CLINICAL TRIAL: NCT02689310
Title: Leptospermum Scoparium Honey and Wound Care for Pressure Ulcers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patients recruited. Study didn't get off the ground. PI left.
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Honey & Wound Care
Record Dates: First submitted 2016-02-08; First posted 2016-02-23 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Pressure Ulcers
Keywords: Wound Care; Medical Grade Honey; Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Care - Stage III Pressure Ulcers (Other): Patients with a stage III pressure ulcer who are randomized into this arm will be given standard treatment (hydrogel, collegense, and silver alginate dressings).
  Interventions: Other: Standard of Care Treatment
- Honey Treatment - Stage III Pressure Ulcers (Experimental): Patients with a stage III pressure ulcer who are randomized into this treatment arm will be given leptospermum scoparium honey dressings for treatment of their wound.
  Interventions: Other: Leptospermum scoparium honey
- Standard Care - Stage IV Pressure Ulcers (Other): Patients with a stage IV pressure ulcer who are randomized into this arm will be given standard treatment (hydrogel, collegense, and silver alginate dressings).
  Interventions: Other: Standard of Care Treatment
- Honey Treatment - Stage IV Pressure Ulcers (Experimental): Patients with a stage IV pressure ulcer who are randomized into this treatment arm will be given leptospermum scoparium honey dressings for treatment of their wound.
  Interventions: Other: Leptospermum scoparium honey

INTERVENTIONS:
Other: Leptospermum scoparium honey — No information available- PI left- study being withdrawn.
  Arms: Honey Treatment - Stage III Pressure Ulcers; Honey Treatment - Stage IV Pressure Ulcers
Other: Standard of Care Treatment — No information available- PI left- study being withdrawn.
  Arms: Standard Care - Stage III Pressure Ulcers; Standard Care - Stage IV Pressure Ulcers

SUMMARY:
The investigators hypothesize that the use of leptospermum scoparium honey as a type of dressing and/or debridement agent on stage III or IV pressure ulcers has an increased efficacy and safety compared to the current treatment protocol that includes the use of hydrogel/Vaseline, collagenase, and silver alginate dressings as the standard of care. Utilizing a non-inferiority trial, it is expected that the use of leptospermum scoparium as a treatment for Stage III and Stage IV pressure ulcers will not be inferior to the comparison treatment of standard of care wound dressings. Moreover, this research design will enable the research team to determine if the honey based dressings are equivalent to or superior to the comparison treatment.

Therefore, the investigators specific study objectives are as follows:

1. Primary Objectives: Determine if the use of honey as an alternative treatment will reduce site inflammation/irritation and pain associated with pressure ulcers compared to the standard treatment options. Specifically, the investigators will monitor patient PUSH scores, Braden Risk Scale scores, granulation and/or epithelial tissue progression, length of time to heal, patient pain assessments via the Wong Baker Face or Numeric Scale, wound odors, and incidence of adverse events (measured by allergies, stinging sensations, bacterial infections that warrant antibiotic intervention, etc.).
2. Secondary Objective: Patients in the honey treatment group will have lower costs per healed ulcer than patients in the standard collagenase treatment group.

DETAILED DESCRIPTION:
Design: Non-inferiority Trial. This design is intended to demonstrate that Leptospermum scoparium Honey treatment is no worse than the standard treatment for pressure ulcers.

Data Collection Procedures:

Members of the research team will administer all wound care treatments on all of the patients in this research project. After initial evaluation and documentation of the presence of pressure ulcers, patients with Stage III and Stage IV ulcers are randomized into the two groups; treatment and control. Patients that develop nosocomial Stage III and Stage IV pressure ulcers will also be included in this study and randomly placed into one of the groups. The following protocol will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years old and older)
* Newly admitted patients with a diagnosis Pressure Ulcers (Stages III and IV) or patients who develop nosocomial pressure ulcers Stage III and Stage IV
* Ability to provide written informed consent (either patient or legal personal representative)

Exclusion Criteria:

* Patient/representative refuses to give written informed consent
* Patient diagnosed with terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Total Score on the Pressure Ulcer Scale for Healing (PUSH) Scale | 6 weeks
  Developed by the National Pressure Ulcer Advisory Panel (NPUAP) as a quick and reliable tool to monitor the change in pressure ulcer status over time and has been incorporated as a standard assessment tool in acute care settings.
Odor (scored as no odor, odor on dressing change, odor all the time) | 6 weeks
  Observed by staff and patient, will be scored as no odor, odor on dressing change, odor all the time.
Incidence of adverse events | 6 weeks
Braden Scale assessment | 6 weeks
Irritation | 6 weeks
  Presence or absence of irritation as determined by clinical observation
Inflammation | 6 weeks
  Presence or absence of irritation as determined by clinical observation
Pain | 6 weeks
  Pain in and around pressure ulcer assessed by tenderness to the touch by clinician (recorded as present or absent)

SECONDARY OUTCOMES:
Costs treated per ulcer | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- NYC Health + Hospitals/Coney Island, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided